CLINICAL TRIAL: NCT00531960
Title: A Randomized, Open-label Study Comparing the Anti-tumor Effect of Treatment With Tarceva Plus Avastin Versus Chemotherapy Plus Avastin in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: A Study of Tarceva (Erlotinib) in Combination With Avastin (Bevacizumab) in Patients With Advanced Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO20571
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Bevacizumab

ARMS (2):
- Bevacizumab, Chemotherapy (Active Comparator): Participants received bevacizumab, 15 milligrams (mg) per (/) kilogram (kg), intravenously (IV), on Day 1 of Cycles 1 through 7 until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received 4 to 6 cycles of a standard platinum-containing regimen of chemotherapy: either gemcitabine, 1250 mg/ square meter (m^2), IV, on Days 1 and 8 of Cycles 1 through 4 or 6, and cisplatin 80 mg/m^2, IV, on Day 1 of Cycles 1 through 4 or 6; or paclitaxel, 200 mg/m^2, IV, and carboplatin area under the curve (AUC) 6 mg/ milliliter (ml) multiplied by (*) minute (min) on Day 1 of Cycles 1 through 4 or 6. The chemotherapy regimen and number of cycles was up to the discretion of the investigator.
  Interventions: Drug: Bevacizumab; Drug: Standard platinum-based chemotherapy
- Bevacizumab, Erlotinib (Experimental): Participants received bevacizumab, 15 mg/kg, IV, on Day 1 of Cycles 1 through 7 until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received erlotinib, 150 mg, orally (PO), daily until disease progression, unacceptable toxicity, death, or withdrawal.
  Interventions: Drug: Erlotinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Erlotinib — 150 mg, PO, daily
  Other Names: Tarceva
  Arms: Bevacizumab, Erlotinib
Drug: Bevacizumab — 15 mg/kg, IV, Day 1 of Cycles 1 through 7
  Other Names: Avastin
Drug: Standard platinum-based chemotherapy — At the discretion of the investigator
  Arms: Bevacizumab, Chemotherapy

SUMMARY:
This 2 arm study will compare the efficacy and safety of Tarceva plus Avastin, and chemotherapy plus Avastin, in the first-line treatment of patients with advanced non-small cell lung cancer. Patients will be randomized to receive either Tarceva 150mg p.o. daily plus Avastin 15mg/kg i.v. every 3 weeks, or standard platinum-based chemotherapy (4-6 cycles) plus Avastin. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced (stage IIIb and IV) non-small cell lung cancer;
* measurable disease;
* ECOG PS 0-1.

Exclusion Criteria:

* prior chemotherapy or treatment with another systemic anti-cancer agent;
* radiotherapy within 4 weeks prior to first dose of study treatment;
* CNS metastases;
* other malignancies in past 5 years, except for adequately treated cancer in situ of the cervix, basal or squamous cell skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- Australia (2):
  - East Bentleigh, Victoria
  - Geelong, Victoria
- Leuven, Belgium
- France (7):
  - Bayonne
  - Dijon
  - Le Mans
  - Marseille
  - Paris
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Italy (4):
  - Aviano, Friuli Venezia Giulia
  - Milan, Lombardy
  - Ancona, The Marches
  - Lido di Camaiore, Tuscany
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (7):
  - 's-Hertogenbosch
  - Amsterdam
  - Eindhoven
  - Groningen
  - Heerlen
  - Maastricht
  - Rotterdam
- Poland (3):
  - Lodz
  - Lublin
  - Otwock
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Timișoara
- Singapore, Singapore
- South Korea (6):
  - Bundang City
  - Daegu
  - Gyeonggi-do
  - Incheon
  - Seoul
  - Suwon
- Spain (6):
  - Alicante, Alicante
  - Barcelona, Barcelona
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Tainan
  - Taipei
- United Kingdom (3):
  - Dudley
  - Guildford
  - Manchester

REFERENCES:
- [Derived] Ciuleanu T, Tsai CM, Tsao CJ, Milanowski J, Amoroso D, Heo DS, Groen HJ, Szczesna A, Chung CY, Chao TY, Middleton G, Zeaiter A, Klingelschmitt G, Klughammer B, Thatcher N. A phase II study of erlotinib in combination with bevacizumab versus chemotherapy plus bevacizumab in the first-line treatment of advanced non-squamous non-small cell lung cancer. Lung Cancer. 2013 Nov;82(2):276-81. doi: 10.1016/j.lungcan.2013.08.002. Epub 2013 Aug 13. PMID 23992877

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Plus (+) Chemotherapy: Participants received bevacizumab 15 milligrams per kilogram (mg/kg), intravenously (IV), on Day 1 of Cycles 1 through 7 (21 day cycles) until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received a maximum of up to 6 cycles (12-18 weeks) with EITHER a gemicitabine/cisplatin regimen (gemcitabine 1250 milligrams per square meter [mg/m^2], IV, on Days 1 and 8 of up to 6 cycles of 21 days, and cisplatin 80 mg/m^2, IV, on Day 1 of up to 6 cycles of 21 days); OR a carboplatin/paclitaxel regimen (paclitaxel 200 mg/m^2, IV, followed by carboplatin 6 milligrams per milliliter multiplied by minute [mg/mL*min] on Day 1 of up to 6 cycles of 21 days). The chemotherapy regimen and number of cycles was up to the discretion of the investigator.
- Bevacizumab + Erlotinib: Participants received bevacizumab 15 mg/kg, IV, on Day 1 of Cycles 1 through 7 (21 day cycles) until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received erlotinib 150 mg tablets, orally (PO), daily until disease progression, unacceptable toxicity, death, or withdrawal.
Period: Overall Study
Arm/Group | Bevacizumab Plus (+) Chemotherapy | Bevacizumab + Erlotinib
Started | 61 | 63
Completed | 0 | 0
Not Completed | 61 | 63
Not completed — Adverse Event | 5 | 4
Not completed — Death | 3 | 2
Not completed — Lack of Efficacy | 42 | 41
Not completed — Violation of Selection Criteria | 2 | 0
Not completed — Refused Treatment | 5 | 6
Not completed — Other | 4 | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all randomized participants.
Groups:
- Bevacizumab + Chemotherapy: Participants received bevacizumab 15 mg/kg, IV, on Day 1 of Cycles 1 through 7 (21 day cycles) until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received a maximum of up to 6 cycles (12-18 weeks) with EITHER a gemicitabine/cisplatin regimen (gemcitabine 1250 mg/m^2, IV, on Days 1 and 8 of up to 6 cycles of 21 days, and cisplatin 80 mg/m^2, IV, on Day 1 of up to 6 cycles of 21 days); OR a carboplatin/paclitaxel regimen (paclitaxel 200 mg/m^2, IV, followed by carboplatin 6 mg/mL*min on Day 1 of up to 6 cycles of 21 days). The chemotherapy regimen and number of cycles was up to the discretion of the investigator.
- Bevacizumab + Erlotinib: Participants received bevacizumab 15 mg/kg, IV, on Day 1 of Cycles 1 through 7 (21 day cycles) until disease progression, unacceptable toxicity, death, or withdrawal. Participants also received erlotinib 150 mg tablets, PO, daily until disease progression, unacceptable toxicity, death, or withdrawal.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib | Total
Number analyzed (Participants) | 61 | 63 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (9.55) | 61.0 (10.94) | 59.53 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Progression-free survival (PFS) was defined as the time from randomization to disease progression or death, from any cause. Progressive disease (PD) was defined according to Response Criteria in Solid Tumors (RECIST) version (V) 1.0. For target lesions (TLs), progressive disease (PD) was defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded since the start of treatment. For non-target lesions (NTLs), PD was defined as unequivocal progression of existing NTLs. Participants were censored at the date of last post-baseline (BL) tumor assessment where non-progression was documented. If no post-BL tumor assessment was available, the participant was censored at date of randomization.
Time Frame: Screening, end of every 2nd cycle through Cycle 8 (21-day cycles), and every 12 weeks thereafter until the end of study and final analysis up to a maximum of 42 months.
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 61 | 63
percentage of participants | 72.1 | 76.2

2. Primary Outcome: PFS
Description: The median time, in weeks, from randomization to PFS event. Participants were censored at the date of last post-BL tumor assessment where non-progression was documented. If no post-BL tumor assessment was available, the participant was censored at date of randomization. PFS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 1
Population: FAS; only participants with an event (disease progression or death) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 44 | 48
weeks | 34.6 [25.0 to 42.4] | 23.4 [17.4 to 45.1]
Statistical Analysis 1: Comparison: Bevacizumab + Chemotherapy vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.8060, Log Rank; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.70 to 1.59]

3. Secondary Outcome: Percentage of Participants Who Died
Description: Overall survival (OS) was defined as the time from randomization to the date of death, due to any cause. Participants were censored at final analysis at the date the participant was last known to be alive.
Time Frame: Screening, Days 1, 8, and 21 of Cycles 1-8 (21-day cycles), and every 12 weeks thereafter until the end of study and final analysis up to a maximum of 42 months.
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 61 | 63
percentage of participants | 45.9 | 52.4

4. Secondary Outcome: OS
Description: The median time, in months, from randomization to OS event. Participants were censored at final analysis at the date the participant was last known to be alive.
Time Frame: as for outcome 3
Population: FAS; only participants who died were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 28 | 33
months | NA [12.7 to NA] — The median and upper limit of the 95% confidence interval (CI) could not be calculated due to the large number of censored events. | 16.4 [11.0 to NA] — The upper limit of the 95% CI could not be calculated due to the large number of censored events.
Statistical Analysis 1: Comparison: Bevacizumab + Chemotherapy vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.4063, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.75 to 2.05]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST V 1.0
Description: BOR was defined as the best response recorded from randomization until disease progression/recurrence or death, taking as reference for PD the smallest measurement (nadir) recorded since treatment started. Assignment of PR of CR required confirmation of tumor measurement changes by repeat assessments performed no less than 4 weeks after criteria for response was first met. For TLs, CR was defined as the disappearance of all TLs; and PR was defined as at least a 30% decrease in the SLD of the TLs, taking BL SLD as reference. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. The 95% CI for one sample binomial was calculated using the Pearson-Clopper method.
Time Frame: as for outcome 1
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 61 | 63
percentage of participants | 44.3 [31.5 to 57.6] | 27.0 [16.6 to 39.7]
Statistical Analysis 1: Comparison: Bevacizumab + Chemotherapy vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.0444, Chi-squared; Difference in Response Rates = -17.28, 95% CI 2-sided [-34.8 to 0.3] — The 95% CI for the difference of 2 rates was determined by using the Hauck-Anderson method

6. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST V 1.0
Description: Disease control was defined as a BOR of CR, PR, or SD according to RECIST V 1.0 for at least 4 weeks at any time during randomized treatment or disease stabilization, after study entry. Participants without a post-BL assessment of response were considered as having no disease control. The 95% CI for the one sample binomial was calculated using the Pearson-Clopper method.
Time Frame: Screening, end of every 2nd cycle through Cycle 8 (21-day cycles), and every 12 weeks thereafter until the end of study and final analysis, 12 months after the last participant's 1st visit
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Number analyzed (Participants) | 61 | 63
percentage of participants | 85.2 [73.8 to 93.0] | 73.0 [60.3 to 83.4]
Statistical Analysis 1: Comparison: Bevacizumab + Chemotherapy vs Bevacizumab + Erlotinib; Test type: Superiority or Other; p = 0.0944, Chi-squared; Difference in Disease Control Rates = -12.2, 95% CI 2-sided [-27.3 to 2.8] — The 95% CI for the difference in disease control was determined using the Hauck-Anderson method

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious AEs (SAEs) were reported from Screening through Day 84. Unrelated events were reported up to 28 days after last study drug treatment, related events were reported until resolution or stabilization
Description: All participants who received at least 1 dose of the study treatment and had at least 1 safety follow-up, whether withdrawn prematurely or not, were included in the safety analysis population.
Arm/Group | Bevacizumab + Chemotherapy | Bevacizumab + Erlotinib
Serious Adverse Events (participants affected / at risk) | 22/60 | 17/63
Other Adverse Events (participants affected / at risk) | 58/60 | 60/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=60) | Bevacizumab + Erlotinib (N=63)
Pneumonia (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Chemotherapy (N=60) | Bevacizumab + Erlotinib (N=63)
Nausea (Gastrointestinal disorders) | 37 | 12
Diarrhoea (Gastrointestinal disorders) | 15 | 27
Vomiting (Gastrointestinal disorders) | 23 | 5
Constipation (Gastrointestinal disorders) | 12 | 7
Stomatitis (Gastrointestinal disorders) | 8 | 9
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 39
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Neutropenia (Blood and lymphatic system disorders) | 24 | 0
Anaemia (Blood and lymphatic system disorders) | 18 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 1
Leukopenia (Blood and lymphatic system disorders) | 17 | 0
Asthenia (General disorders) | 13 | 7
Fatigue (General disorders) | 19 | 14
Mucosal inflammation (General disorders) | 4 | 5
Hypertension (Vascular disorders) | 14 | 19
Headache (Nervous system disorders) | 7 | 12
Neuropathy peripheral (Nervous system disorders) | 10 | 1
Paronychia (Infections and infestations) | 1 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Insomnia (Psychiatric disorders) | 7 | 8
Proteinuria (Renal and urinary disorders) | 9 | 12
Gingival bleeding (Gastrointestinal disorders) | 5 | 3
Toothache (Gastrointestinal disorders) | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1
Periodontitis (Gastrointestinal disorders) | 2 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oral pruritus (Gastrointestinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Chest pain (General disorders) | 6 | 6
Chest discomfort (General disorders) | 4 | 5
Pyrexia (General disorders) | 3 | 6
Pain (General disorders) | 0 | 4
Oedema (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 1
Chills (General disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 2
Axillary pain (General disorders) | 0 | 1
Discomfort (General disorders) | 1 | 0
Feeling cold (General disorders) | 0 | 1
Hunger (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Xerosis (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Vision blurred (Eye disorders) | 3 | 2
Blepharitis (Eye disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 2
Diplopia (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 23 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 4
Paraesthesia (Nervous system disorders) | 5 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Ageusia (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 6
Nasopharyngitis (Infections and infestations) | 4 | 4
Bronchitis (Infections and infestations) | 0 | 3
Folliculitis (Infections and infestations) | 0 | 3
Catheter site infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 2
Aortic thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Weight decreased (Investigations) | 4 | 3
Alanine aminotransferase increased (Investigations) | 1 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood creatinine increased (Investigations) | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 2 | 0
Weight increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Lymphocyte count increased (Investigations) | 1 | 0
Monocyte count increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.